CLINICAL TRIAL: NCT04862078
Title: Shared Decision Making in Follow-up Imaging Surveillance for Distant Metastasis in Treated Breast Cancer Patients [SMART-FU]: A Prospective, Single-institution, Randomized Pragmatic Trial
Brief Title: Shared Decision Making in Surveillance for Distant Metastasis in Breast Cancer
Acronym: SMART-FU
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hyeong-Gon Moon, Medical doctor, Clinical Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2012-090-1182
Record Dates: First submitted 2021-04-18; First posted 2021-04-27 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer; Survivorship; Quality of Life
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shared decision making group (Experimental): The Study arm - shared decision making when deciding surveillance strategy
  Interventions: Diagnostic Test: Shared decision making
- Usual surveillance group (Other): The control arm - surveillance with usual care
  Interventions: Diagnostic Test: Usual care

INTERVENTIONS:
Diagnostic Test: Shared decision making — Shared decision making and decide surveillance strategy between "standard follow-up according to the institutional practice and decide what to do advanced imagings for surveillance" and "guideline-based surveillance"
  Arms: Shared decision making group
Diagnostic Test: Usual care — standard follow-up according to the institutional practice
  Arms: Usual surveillance group

SUMMARY:
In this study, clinical impacts of shared decision making between physicians and patients in strategy of surveillance for asymptomatic patients who ended the primary treatments on quality of life would be investigated

DETAILED DESCRIPTION:
[Background]

1. Shared decision making between patients and physicians when breast cancer patients encounter decision making in the initial treatment process has already been included in the recommendations for breast cancer treatment in each country. However, in the follow-up stage using various imaging tests after the initial breast cancer treatment, the evidence of decision making is very poor and the patient who understands this well and actively participates in the process of deciding the follow-up strategy are almost none.
2. Major guidelines including NCCN, ASCO and ESMO recommend surveillance with routine imaging such as sonography and mammography, and does not recommend advanced imaging tests for asymptomatic patients. These guidelines are based on two prospective randomized trials conducted in 1994. Despite many international medical recommendations, many institutions around the world are increasingly using distant metastasis tests in belief of improving the survival rate through early detection of distant metastasis and of improving the emotional stability of doctors and patients.
3. In this study, clinical impacts of shared decision making in strategy of surveillance for asymptomatic patients on quality of life would be investigated by prospective randomized pragmatic trial. Additionally, oncological results would be analyzed and real world data of patients preference would be gathered

[Study design] Prospective, single-institutional, randomized pragmatic trial

[Statistical considerations] With 5% significance level and 90% power, 132 patients are needed in each group. Assuming a 28% drop out rate, 368 patients need to be recruited.

[Randomizations] Web-based randomization would be conducted stratified to subtypes.

[Objectives]

1. Primary objective

   - QoL (when enrollment, after 1 and 2 year - FACT-B score)
2. Secondary objectives

   * Depression - anxiety scale (HADS score)
   * Recurrence-free survival
   * Patients' preference for surveillance in SDM group
   * Cross over rate in SDM group

ELIGIBILITY:
Inclusion Criteria:

* Women between 20-70 years
* Invasive unilateral breast carcinoma with histological confirmation
* History of invasive breast cancer
* TMN stage I-II according to AJCC 7th
* Histologically or radiologically no suspicion of distant metastases
* Performance status corresponding to ECOG grade 0-2
* No psychological and geographical restriction in follow-up
* Written informed consent

Exclusion Criteria:

* History of any cancer in the previous 5 years
* Bilateral breast cancer
* Male breast cancer
* Patients who are planning for surveillance in other institutions
* Unable to understand and fill out questionnaires

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Estimated)
Dates: Start 2021-07-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of life (QoL), Depression-anxiety scale | At the point of enrollment
  Evaluated QoL with Functional Assessment of Cancer Therapy - Breast (FACT-B) questionnaire
Quality of life (QoL), Depression-anxiety scale | After 6 month of enrollment
  Evaluated QoL with Functional Assessment of Cancer Therapy - Breast (FACT-B) questionnaire
Quality of life (QoL), Depression-anxiety scale | After 1 year of enrollment
  Evaluated QoL with Functional Assessment of Cancer Therapy - Breast (FACT-B) questionnaire
Quality of life (QoL), Depression-anxiety scale | After 2 year of enrollment
  Evaluated QoL with Functional Assessment of Cancer Therapy - Breast (FACT-B) questionnaire

SECONDARY OUTCOMES:
Rate of patients who choose guideline-dependent surveillance rather than advanced imaging-dependent in SDM group | 6 month
  Rate of patients who choose guideline-dependent surveillance in SDM group (Patients' preference for surveillance)
Cross over rate in SDM group | 2 years
  Evaluated Patients' cross-over rate in SDM group

CONTACTS AND LOCATIONS:
Overall Officials: Hyeong-Gon Moon, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea